CLINICAL TRIAL: NCT05363345
Title: Randomized Trial of the Removal Ability With Vortic Catch V Basket Catheter Versus Ordinary Basket Catheter for Bile Duct Stones
Brief Title: Comparison of Vortic Catch V Basket Catheter and Ordinary Basket Catheter for the Removal of Bile Duct Stones
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Akira Horiuchi (Other)
Responsible Party: Sponsor-Investigator, Akira Horiuchi, Chief of Digestive Disease Center, Showa Inan General Hospital
Organization: Showa Inan General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Vortic Catch V
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Randomized Study

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vortic Catch V basket catheter (Experimental): Common bile duct stones (≧ 10 mm) are removed by using Vortic Catch V basket catheter following endoscopic papillary large balloon dilation.
  Interventions: Device: bile duct stone removal
- ordinary basket catheter (Active Comparator): Common bile duct stones (≧ 10 mm) are removed by using ordinary basket catheter following endoscopic papillary large balloon dilation.
  Interventions: Device: bile duct stone removal

INTERVENTIONS:
Device: bile duct stone removal — Common bile duct stones (≧ 10 mm) are removed by using Vortic Catch V basket catheter or ordinary basket catheter following endoscopic papillary large balloon dilation.

SUMMARY:
Investigators will perform randomized trial of the removal ability with Vortic Catch V basket catheter versus ordinary basket catheter for bile duct stones (≧ 10 mm).

ELIGIBILITY:
Inclusion Criteria:

* patients with suspected of having, or known to have, common bile duct stones (≧ 10 mm)
* endoscopic papillary balloon dilation (EPLBD) was performed.

Exclusion Criteria:

* septic shock
* coagulopathy (international normalized ratio 1.3, partial thromboplastin time greater than twice that of control),
* <platelet count 50,000 / L
* suspected or confirmed malignancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-02-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of stones cleared | Procedure time
  Percentage of stones cleared is evaluated after the completion of procedure.

SECONDARY OUTCOMES:
Total procedural time | Procedure time
  Total procedure time is measured.
the number of adverse events | Procedure time
  Adverse events are evaluated after the completion of procedure.
the numbers of morbidities and mortality | 30 days
  Morbidities and mortality is evaluated within 30 days after the completion of procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Showa Inan General hospital, Komagane, Nagano, Japan

IPD SHARING:
Plan to Share IPD: No